CLINICAL TRIAL: NCT04127656
Title: Symptom Changes in Infants Fed an Amino Acid-based Formula
Brief Title: Infants Fed an Amino Acid-based Formula
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL28
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amino Acid-Based Experimental Study Formula (Experimental): Single-Arm Study
  Interventions: Other: Amino Acid-Based Experimental Study Formula

INTERVENTIONS:
Other: Amino Acid-Based Experimental Study Formula — Amino Acid-Based Formula; fed ad libitum

SUMMARY:
To observe the effects of an amino acid-based formula on symptoms associated with food allergies in infants.

ELIGIBILITY:
Inclusion Criteria:

* Subject is judged to be in good health as determined from subject's medical history
* Subject is from a full-term birth with a gestational age of 37-42 weeks
* Subject's birth weight was ≥ 2490 g (~5 lbs. 8 oz.)
* Subject has been documented to have CMPA and/or multiple food allergies, FPIES or gastrointestinal eosinophilic disorders.
* Subject is experiencing persistent feeding intolerance symptoms including any of the following: regurgitation/vomiting associated with feeding (within 1 hour), constipation, diarrhoea, hematochezia (blood in the stool), crying, gassiness (wind), and/or skin rash/eczema.
* Parent(s) confirm their intention to feed their infant study product during the study period.
* Parent(s) confirm their intention not to administer vitamin or mineral supplements to their infant from enrolment through the duration of the study, unless instructed otherwise by their healthcare professional.
* Infant using medications (OTC medications for gas [wind]), home remedies (such as juice for constipation), herbal preparations, prebiotics, probiotics or rehydration fluids that might affect Gl tolerance may not be enrolled unless the parent agrees to discontinue the use of these agents prior to enrolment or a healthcare professional recommends their continued use.
* Subject's parent(s) has voluntarily signed and dated an ICF, approved by an IEC/IRB and provided applicable privacy regulation authorisation prior to any participation in the study.

Exclusion Criteria:

* Subject is receiving steroids or antibiotics
* Subject is tube-fed
* Subject has received an amino acid-based formula
* Subject has been diagnosed with: Short bowel syndrome, Inflammatory bowel disease, Pancreatic disease, Protein maldigestion (malnutrition), Mast cell disorder
* Subject is participating in another study that has not been approved as a concomitant study by AN

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Food Allergy Symptom Improvement | Baseline to Day 28
  Parent Completed Symptom Diary

SECONDARY OUTCOMES:
Time to Symptom Resolution or Reduction | Baseline to Day 28
  Parent Completed Symptom Diary
Change in Length | Baseline to Day 28
  Length-for-age z scores
Change in Weight | Baseline to Day 28
  Weight-for-age z scores
Study Formula Intake | Baseline to Day 28
  Parent Completed Intake Diary

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kajzer, MS, RD, LD, Study Chair — Abbott Nutrition
Locations (3):
- United Kingdom (3):
  - The Adam Practice, Poole
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Royal London Hospital, Whitechapel

IPD SHARING:
Plan to Share IPD: No